CLINICAL TRIAL: NCT00059384
Title: Concentration-Controlled Antiretroviral Therapy in Persons Experiencing Persistent Viremia
Brief Title: Alternative Dosing Strategy for Anti-HIV Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R01AI033835-08A1 (NIH); 5M01RR000400-340420; 3M01RR000400-34S1A20420ú
Record Dates: First submitted 2003-04-23; First posted 2003-04-24 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: Treatment experienced; Therapeutic Drug Monitoring
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Concentration-controlled therapy

SUMMARY:
Anti-HIV drugs are usually given to patients at fixed, standardized doses. This study will investigate alternative ways of dosing anti-HIV drugs to improve viral control.

Study hypothesis: The optimal dosage regimen required to obtain the maximum benefit from antiretroviral therapy is achieved with strategies that control for pharmacokinetic and pharmacodynamic variability among patients.

DETAILED DESCRIPTION:
While optimism for the benefits of antiretroviral therapy remain justified, the response to therapy varies widely. This variability arises because of differences among patients in virologic, immunologic, behavioral, and pharmacologic factors, all of which impact therapeutic success.

Antiretroviral agents are presently administered to adults in standard fixed doses. However, the same dose does not produce the same systemic and intracellular concentrations in all patients. Recent research has shown that adjusting the doses of antiretroviral agents to achieve target concentrations in plasma is associated with an improved anti-HIV response compared with standard dose therapy. This study will extend the paradigm of concentration-controlled therapy to develop intensified pharmacologic regimens for patients experiencing persistent viremia while receiving antiretroviral therapy.

Two approaches will be investigated: 1) a regimen that targets concentrations of each antiretroviral drug between the 50th and 75th percentile of expected concentrations in adults; and 2) a novel regimen in which the target concentrations are based upon a desired ratio between phenotypic drug susceptibility (IC90) and the concentrations of pharmacologically active moieties, specifically intracellular nucleoside triphosphates and unbound protease and nonnucleoside inhibitors.

Participants will be randomized to either one of the investigational approaches (Cohort II) or to a control group receiving standard dose therapy (Cohort I). There are two study visits in the first month; after the first month, study visits are scheduled monthly for five additional months. Study visits include laboratory tests of virologic and immunologic parameters, pharmacokinetic sampling, and adherence counseling and monitoring.

ELIGIBILITY:
Inclusion Criteria for Cohort I:

* HIV infected
* Receiving therapy with 3 or more antiretroviral medications and and willing to continue this regimen
* Achieved a greater than 1 log10 reduction in plasma HIV-RNA from baseline within 8 weeks after the start of current therapy
* Current plasma HIV-RNA levels greater than 500 copies/mL and less than 10,000 copies/mL

Inclusion Criteria for Cohort Cohort II:

* HIV infected
* Receiving antiretroviral therapy and have been determined to have had virologic failure
* Will or have been changed to a new antiretroviral regimen (addition of greater than one new antiretroviral agent), but have not received this new regimen for more than 4 weeks as of study entry
* HIV RNA of 2500 copies/mL or greater at screening

Exclusion Criteria:

* Concurrent investigational antiretroviral agent
* Malignancy, including Kaposi's sarcoma, requiring systemic chemotherapy
* Active opportunistic infection requiring therapy within 14 days prior to study entry
* Drug-resistant mutations that necessitate a change in antiretroviral regimen
* Active drug or alcohol use or dependence
* Certain laboratory abnormalities
* Pregnant or breastfeeding
* Known nonadherence with medications and scheduled clinic visits
* Any medical condition that, in the opinion of the investigators, would preclude successful completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Ability of the concentration-controlled strategies to achieve and maintain target concentrations
safety and tolerability of pharmacologic intensification
ability of pharmacologic intensification to achieve and maintain a sustained suppression in plasma HIV RNA

SECONDARY OUTCOMES:
Cross clade neutralizing antibody
cellular immunity

CONTACTS AND LOCATIONS:
Overall Officials: Courtney V. Fletcher, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Denver, Colorado, United States